CLINICAL TRIAL: NCT01985568
Title: Optimal Timing of Exercise Initiation Within a Lifestyle Weight Loss Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-1550; R01DK097266 (NIH)
Record Dates: First submitted 2013-10-24; First posted 2013-11-15 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Obesity
Keywords: Obesity; weight-loss; Physical activity
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Behavioral Therapy (Standard BT) (Active Comparator): Standard BT: This group will follow a traditional model of initiating exercise concurrently with a dietary intervention for weight loss within an 18 month behavioral weight loss program.
  Interventions: Behavioral: Standard BT
- Sequential Behavioral Therapy (Sequential BT) (Experimental): Sequential BT: This group will receive diet and exercise interventions delivered sequentially within an 18 month behavioral weight loss program.
  Interventions: Behavioral: Sequential BT

INTERVENTIONS:
Behavioral: Sequential BT — Both study arms (Standard BT and Sequential BT) will receive an identical 6 month group-based weight loss program, followed by an identical 6 month group-based weight maintenance program, followed by an identical 6 months of weight maintenance phone support. Both groups will also receive an identical 6 month exercise intervention. Groups will differ only in the timing of exercise initiation. Sequential BT will be asked not to begin exercise during months 0-6. They will receive a progressive exercise program and exercise behavior support during months 7-12.
  Arms: Sequential Behavioral Therapy (Sequential BT)
Behavioral: Standard BT — Both study arms (Standard BT and Sequential BT) will receive an identical 6 month group-based weight loss program, followed by an identical 6 month group-based weight maintenance program, followed by an identical 6 months of weight maintenance phone support. Both groups will also receive an identical 6 month exercise intervention. Groups will differ only in the timing of exercise initiation. Standard BT will begin exercise immediately upon starting the 6 month dietary weight loss intervention. They will receive a progressive exercise program and exercise behavior support during months 0-6.
  Arms: Standard Behavioral Therapy (Standard BT)

SUMMARY:
The primary aim of this study is to evaluate the extent to which an exercise intervention timed after diet-induced weight loss (rather than initiated at the same time) improves exercise adherence and long-term weight loss. An 18 month randomized trial will be used to compare two behavioral weight loss programs; standard behavioral therapy (Standard BT) and sequential behavioral therapy (Sequential BT). The Standard BT group will receive a traditional behavioral weight loss program where diet and exercise changes are initiated at the same time. The Sequential BT group will receive a program that focuses solely on dietary changes in the initial 6 months, and then incorporates exercise in the ensuing 6 months. Both groups will be followed for 18 months to assess long-term weight loss. The hypothesis is that delivery of diet and exercise interventions in sequence will result in improved adherence to exercise and weight loss at 18 months when compared to a traditional program in which identical diet and exercise interventions are initiated at the same time. This study could identify a strategy that could aid in the development of more effective obesity treatment programs and help more people achieve and sustain a weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* Body Mass Index 27-42 kilograms/meters squared
* Sedentary: defined as regular exercise of less than 100 minutes per week at moderate intensity or greater during the previous 6 months
* No self-report of acute or chronic disease (heart disease, diabetes, gastrointestinal disorders and orthopedic problems in particular)
* No plans to relocate or for extended travel (more than 1 week) within the next 18 months
* No current tobacco use
* Capable and willing to give informed consent, understand exclusion criteria, and accept the randomized group assignment
* Live or work within 20 minutes of the University of Colorado Anschutz Health and Wellness Center to ensure reasonable ability to comply with requirement to attend group weight loss sessions and supervised exercise sessions. Exceptions can be made at the discretion of the Study Principal Investigator (PI) on a case by case basis for highly motivated subjects.
* For Females

  * Not currently pregnant or lactating
  * Not pregnant within the past 6 months
  * Not planning to become pregnant in the next 18 months
  * Sexually active women of childbearing potential may be enrolled if they have had a tubal ligation or use a reliable means of contraception.

Exclusion Criteria:

* Presence or history of health problems which would affect appetite, food intake, energy metabolism, or ability to optimally participate in the exercise component including: diabetes, cardiovascular disease, peripheral vascular disease, cerebrovascular disease, uncontrolled hypertension, uncontrolled hyper or hypothyroidism, cancer (within the last 5 years, except skin cancer), human immunodeficiency virus (HIV) infection, significant gastrointestinal, pulmonary, renal, musculoskeletal, neurologic, or hematologic disease
* Symptoms suggestive of cardiovascular disease: chest pain, shortness of breath at rest or with mild exertion, syncope
* Abnormal resting electrocardiogram (ECG): serious arrhythmias, including multifocal Premature Ventricular Contractions (PVCs), frequent PVC's (defined as 10 or more per minute), ventricular tachycardia (defined as runs of 3 or more successive PVC's), or sustained atrial tachyarrhythmia; 2nd or 3rd degree A-V block, corrected QT interval > 480 millisecond or other significant conduction defects
* Triglycerides > 400 milligram/deciliter (md/dL) or Low-Density Lipoprotein (LDL) cholesterol > 190 mg/dL
* Use of prescription or over-the-counter medications known to affect appetite, weight, heart rate response to exercise, or energy metabolism
* Use of systemic steroids (other than Oral Contraceptive Pills)
* Use of obesity pharmacotherapeutic agents within the last 6 months
* History of surgical procedure for weight loss
* History of major surgery within the past 3 months
* Current alcohol or substance abuse
* History of clinically diagnosed eating disorders including anorexia nervosa or bulimia
* Current severe depression or history of severe depression within the previous year
* History of other significant psychiatric illness (e.g. psychosis, schizophrenia, mania, bipolar disorder) which in the opinion of the Study MD would interfere with ability to adhere to dietary or exercise interventions
* Currently participating in or planning to participate in any formal weight loss or physical activity programs or clinical trials
* Weight loss or gain of > 5% in past 6 months for any reason except post-partum weight loss
* Participation in a weight loss program using the Colorado Weigh curriculum within the past 3 years (exceptions can be made at the discretion of the study PI on a case-by-case basis).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2013-11; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | Baseline, 3, 6, 9, 12, 15, and 18 months.
  Body weight will be assessed.
Change in Body Composition | Baseline, 6, 12, and 18 months.
  Body composition will be assessed.

SECONDARY OUTCOMES:
Objectively Measured Change in Physical Activity | Baseline, 6, 12, and 18 months.
  Physical activity will be measured with activity monitors.
Change in Maximal Aerobic Capacity | Baseline, 6, 12, and 18 months.
  Maximal aerobic capacity will be measured.
Change in Diet Composition | Baseline, 6, 12, and 18 months.
  Dietary energy intake (calories/day) and fat intake (grams/day) will be measured.
Change in Engagement in Weight Control Eating Behaviors | Baseline, 6, 12, and 18 months.
  Engagement in weight control eating behaviors will be measured with a questionnaire.
Change in Dietary Weight Loss Program Attendance and Adherence | 18 months
  Dietary weight loss program attendance and adherence will be assessed throughout the 18 month program.
Change in Exercise Program Attendance and Adherence | 18 months
  Exercise program attendance and adherence will be assessed throughout the 18 month program.

OTHER OUTCOMES:
Change in Number of Exercise Related Injuries and Adverse Events | 18 months
  Exercise related injuries and adverse events will be assessed throughout the 18 month program.
Change in Mood | Baseline, 6, 12, and 18 months.
  Mood will be assessed with a questionnaire.
Change in Exercise Self-Efficacy | Baseline, 6, 12, and 18 months.
  Exercise self-efficacy will be assessed with a questionnaire.
Change in Diet Self-Efficacy | Baseline, 6, 12, and 18 months.
  Diet self-efficacy will be assessed with a questionnaire.
Change in Beliefs About Exercise Benefits and Barriers | Baseline, 6, 12, and 18 months.
  Beliefs about exercise benefits and barriers will be assessed with a questionnaire.
Change in Motivation to Engage in a Weight Loss Treatment Program | Baseline, 6, 12, and 18 months.
  Motivation for engaging in a weight-loss treatment program will be assessed with a questionnaire.
Change in Motivation to Engage in Exercise | Baseline, 6, 12, and 18 months.
  Motivation to engage in exercise will be assessed with a questionnaire.
Change in Physical Activity Enjoyment | Baseline, 6, 12, and 18 months.
  Physical activity enjoyment will be assessed with a questionnaire.
Change in Dietary Self-Control | Baseline, 6, 12, and 18 months.
  Dietary self-control will be assessed with a questionnaire.
Change in Perceived Effort for Weight Control | Baseline, 6, 12, and 18 months.
  Perceived effort for weight control will be measured with a questionnaire.
Change in Post intervention follow-up | 24 months
  Weight, objectively measured physical activity, and outcome measures #6 and #10-18 will be assessed 6 months after completion of intervention.
Change in Genetic and Epigenetic markers | Baseline
  Baseline genetic and epigenetic biomarkers will be analyzed to determine if they are associated with baseline measures and/or changes in post-intervention measure outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Catenacci, MD, Principal Investigator — University of Colorado Anschutz Health and Wellness Center
Locations (1):
- University of Colorado, Anschutz Health and Wellness Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Creasy SA, Ostendorf DM, Kaizer L, Rosenberg R, Breit MJ, Bessesen DH, Melanson EL, Catenacci VA. Effect of physical activity on changes in weight and aerobic capacity during an 18-month behavioral weight loss intervention. Int J Behav Nutr Phys Act. 2025 May 21;22(1):57. doi: 10.1186/s12966-025-01754-3. PMID 40399945
- [Derived] Creasy SA, Ostendorf DM, Blankenship JM, Grau L, Arbet J, Bessesen DH, Melanson EL, Catenacci VA. Effect of sleep on weight loss and adherence to diet and physical activity recommendations during an 18-month behavioral weight loss intervention. Int J Obes (Lond). 2022 Aug;46(8):1510-1517. doi: 10.1038/s41366-022-01141-z. Epub 2022 May 16. PMID 35577898
- [Derived] Ostendorf DM, Schmiege SJ, Conroy DE, Phelan S, Bryan AD, Catenacci VA. Motivational profiles and change in physical activity during a weight loss intervention: a secondary data analysis. Int J Behav Nutr Phys Act. 2021 Dec 4;18(1):158. doi: 10.1186/s12966-021-01225-5. PMID 34863198
- [Derived] Catenacci VA, Ostendorf DM, Pan Z, Bing K, Wayland LT, Seyoum E, Stauffer BL, Phelan S, Creasy SA, Caldwell AE, Wyatt HR, Bessesen DH, Melanson EL. The Impact of Timing of Exercise Initiation on Weight Loss: An 18-Month Randomized Clinical Trial. Obesity (Silver Spring). 2019 Nov;27(11):1828-1838. doi: 10.1002/oby.22624. Epub 2019 Sep 29. PMID 31565869